CLINICAL TRIAL: NCT04295798
Title: Optimizing Transcranial Direct Current Stimulation (tDCS) to Improve Dual Task Gait and Balance in Older Adults
Brief Title: Optimizing tDCS to Improve Dual Task Gait and Balance
Acronym: OptiStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Brad Manor, Associate Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019-23
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Aging
Keywords: Mobility; Dual Task

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a "within-subject," double-blinded, randomized controlled study comparing the after-effects of single sessions of conventional tDCS, optimized tDCS, and two different sham conditions on dual task performance in men and women aged 65-85 years with poor baseline dual task performance. Participants will complete an optional structural brain MRI. They will then complete four visits during which they will receive one of the four interventions in random order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study personnel administering tDCS and the participants will not be aware of tDCS intervention arm assignment. The investigators will ensure such double-blinding by programming the tDCS software with intervention-specific stimulation codes, as supplied by personnel uninvolved in data collection, prior to study initiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional tDCS (Experimental): One 20-minute session of active tDCS using two 35 cm2 sponge electrodes targeting the left dlPFC.
  Interventions: Device: Conventional tDCS
- Optimized tDCS (Experimental): One 20-minute session of active tDCS using eight gel electrodes with placement and current parameters optimized to the cohort targeting the left dlPFC.
  Interventions: Device: Optimized tDCS
- Conventional sham (Sham Comparator): One 20-minute session of inactive sham tDCS delivered via two sponge electrodes for a short period of time before it is ramped down to zero for the remainder of the session.
  Interventions: Device: Conventional Sham
- Optimized Sham (Sham Comparator): One 20-minute session of active sham in which the Stimweaver optimization algorithm will be used with the objective of creating a null electric field on the target left dlPFC with the constraint that some gel electrodes deliver low-level currents that still induce cutaneous sensations.
  Interventions: Device: Optimized Sham

INTERVENTIONS:
Device: Conventional tDCS — The anode will be placed over F3 and the cathode over the contralateral supraorbital margin. At the beginning of stimulation, the current will be increased from 0.1 mA, in 0.1 mA increments over 60 seconds, up to a maximum of 1.8 mA. At the end of each session, current will be automatically ramped down to 0.0 mA over a 60 second period.
  Arms: Conventional tDCS
Device: Optimized tDCS — This intervention will utilize eight gel electrodes with placement and current parameters optimized to the cohort, with the goal of generating an average nE over the left dlPFC of the same size as the one delivered by a conventional montage using sponges. The direct current delivered by any one electrode will however never exceed 2.0 mA; the total amount of current from all electrodes will not exceed 4 mA. Each 20- minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Arms: Optimized tDCS
Device: Conventional Sham — Conventional sham will be used to maximize blinding of conventional sponge-based stimulation. The same sponge placement, ramp-up procedure, and session duration described above will be used; however, current will be automatically ramped down 60 seconds after ramp-up.
  Arms: Conventional sham
Device: Optimized Sham — An active sham will be used in which very low-level currents (0.5 mA max) are transferred between the same electrodes used in the active condition throughout the entire 20-minute session. This intervention will be optimized to deliver currents designed to not significantly influence their cortical tissue, but still mimic the cutaneous sensations induced by tDCS. We have shown that this active sham effectively blinds participants and operators to stimulation condition and does not affect functional outcomes.
  Arms: Optimized Sham

SUMMARY:
The objective of this study is to determine the acute effects of single sessions of optimized tDCS, conventional tDCS, and sham stimulation on dual task standing and walking in older adults who are free of overt disease yet who present with poor baseline dual task performance.

DETAILED DESCRIPTION:
Standing and walking are almost always completed in unison with other cognitive tasks such as talking, reading or making decisions. The ability to perform this important type of "dual tasking" is critical to daily activities and dependent upon one's capacity to effectively activate appropriate brain networks that include the left dorsolateral prefrontal cortex (dlPFC). Transcranial direct current stimulation (tDCS) is a safe, noninvasive technology that can selectively modulate brain excitability (i.e., the likelihood of activation) by passing low-level currents between electrodes placed upon the scalp. We have demonstrated through a series of studies that a single, 20-minute exposure of 'conventional' tDCS targeting the left dlPFC-administered via two large sponge electrodes-reduces dual task costs to metrics of standing postural control and gait, when tested immediately following stimulation. Still, we and others have also observed relatively high between-subject variability in the effects of this conventional bipolar form of tDCS. We contend that this variability in effectiveness arises in part from relatively diffuse and unspecific current flow when using large sponge electrodes, in combination with individual variability in head and brain anatomy that significantly alters current flow and the generated electric field in the target brain region.

In this project, we will 1) apply recent advances in tDCS modeling and administration to model the electric fields generated by conventional tDCS in older adults using their individual structural brain MRIs, and 2) develop and test an multi-channel tDCS montage designed to optimize current flow to the left dlPFC (i.e., 'optimized' tDCS). Our Specific Aim is to examine the immediate after-effects of conventional tDCS, optimized tDCS, and sham stimulation on dual task standing and walking in older adults. Our study population will be older men and women without overt disease or illness, yet with poor baseline dual task performance defined as a dual task cost (i.e., reduction) to gait speed of at least 10% induced by simultaneously performing a serial subtraction task when walking. We hypothesize that across participants, the effect of conventional tDCS on dual task standing and walking performance will correlate with a specific component of the electric field generated over the left dlPFC target. We also hypothesize that optimized tDCS will induce A) greater effects on dual task standing and walking performance as compared to conventional tDCS and sham stimulation, and B) these effects will be more consistent across individuals as compared to conventional tDCS.

This project will provide important insights into tDCS "dosage" that will enable us and many other researchers to better understand, control, and optimize this form of noninvasive brain stimulation to individual head and brain anatomy. It is also expected to demonstrate that optimized tDCS, as compared to the conventional approach, significantly improves the size and consistency of observed benefits to dual task standing and walking in vulnerable older adults.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65-85 years
* Poor dual task performance, defined as a preferred gait speed that is >10% slower when walking and simultaneously performing verbalized serial subtractions (i.e., dual tasking), as compared to walking normally (i.e. single tasking)

Exclusion Criteria:

* Unwillingness to cooperate or participate in the study protocol
* An inability to walk or stand for 30 continuous seconds without an assistive device
* A diagnosis of a gait disorder, Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, previous stroke or other neurodegenerative disorder
* Self-report of acute illness, injury or other unstable medical condition; Any report of severe lower-extremity arthritis or pain, physician-diagnosis of peripheral neuropathy, or other peripheral neuromuscular disease that may confound the effects of tDCS on gait or postural control
* Use of antipsychotics, anti-seizure, benzodiazepines, or other neuroactive medications
* Severe depression defined by a Geriatric Depression Scale score greater than 11;
* Any report or physician-diagnosis of schizophrenia, bipolar disorder or other psychiatric illness
* Contraindications to MRI or tDCS, including reported seizure within the past two years, use of neuro-active drugs, the risk of metal objects anywhere in the body, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Marcus Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, physiologic, and brain imaging data, from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.

RESULTS

PARTICIPANT FLOW:
Groups:
- Crossover tDCS: On each visit, participants were randomly assigned to receive one of four different 20-minute tDCS interventions: Conventional tDCS, Optimized tDCS, Conventional Sham, and Optimized Sham.
Period: Overall Study
Arm/Group | Crossover tDCS
Started | 29
Conventional tDCS | 29
Optimized tDCS | 29
Conventional Sham | 29
Optimized Sham | 28
Completed | 28
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Four Interventions in a Cross-over Design: Each subject participated in four sessions of interventions in different days. Conventional tDCS: One 20-minute session of active transcranial direct current stimulation (tDCS) using large sponge electrodes targeting the left dorsolateral prefrontal cortex.
  Optimized tDCS: One 20-minute session of active transcranial direct current stimulation (tDCS) using eight gel electrodes with placement and current parameters optimized to the cohort targeting the left dorsolateral prefrontal cortex.
  Conventional Sham: One 20-minute session of inactive sham in which tDCS will be delivered via sponge electrodes for a short period of time before it is ramped down to zero for the remainder of the session.
  Optimized Sham: One 20-minute session of active sham in which the Stimweaver optimization algorithm will be used with the objective of creating a null electric field on the target (left dlPFC) with the constraint that some gel electrodes deliver low-level currents that still induce cutaneous sensations.
Arm/Group | Four Interventions in a Cross-over Design
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.64 (4.70)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Dual Task Cost to Gait Speed From Baseline to Immediately Post Intervention
Description: Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer, on the low back and feet to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed pre and post tDCS. Two at a preferred speed while walking quietly (single task), two at a preferred speed while performing a cognitive task (dual task) and two fast walking trials. The cognitive task during the dual task condition was verbalized serial subtractions of 3's from a random three-digit number. The absolute change was then calculated using post-intervention dual task cost minus baseline dual task cost. The outcome was calculated by averaging the dual task costs of the four trials. Negative numbers demonstrate lower (i.e., better) dual task cost post intervention. The preferred Unit of Measure is unitless.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Optimized tDCS: One 20-minute session of active tDCS using two 35 cm2 sponge electrodes targeting the left dlPFC.
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
unitless | -2.29 (4.35) | -3.88 (2.77) | 0.06 (4.71) | -0.10 (3.21)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task cost to gait speed from baseline to immediately post intervention; Test type: Equivalence — Model effects included stimulation condition (i.e., gel-tDCS, sponge-tDCS, gel-sham and sponge-sham), time (pre-, post-stimulation), and their interaction. Previous studies showed age, sex, and BMI were associated with one or more metrics of standing or walking and were therefore included as covariates. Tukey's post-hoc testing was used to compare factor means of significant models; p = 0.02, ANOVA

2. Primary Outcome: Absolute Change in Dual Task Cost to Standing Postural Sway Speed From Baseline to Immediately Post Intervention
Description: Postural sway speed was assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during six, 45-second trials of standing with eyes open (single task), eyes closed, or performing a cognitive task (dual task standing) on a stationary force platform (Kistler, Amherst, NY). The cognitive task was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change was then calculated using post-intervention dual task cost minus baseline dual task cost. The outcome was obtained by averaging the dual task costs of the four trials. Negative numbers demonstrate lower (i.e., better) dual task cost post intervention. The preferred Unit of Measure is unitless.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
unitless | -7.66 (10.38) | -5.97 (11.03) | 26.88 (9.83) | 5.06 (11.03)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task cost to standing postural sway speed from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, ANOVA

3. Secondary Outcome: Absolute Change in Dual Task Cost to Stride Time Variability From Baseline to Immediately Post Intervention
Description: Stride time variability is a measure of how consistent limb movements are during walking and is expressed as the coefficient of variation. Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed. Two at a preferred speed while walking quietly (single task), two at a preferred speed while performing a cognitive task (dual task) and two fast walking trials. The cognitive task during the dual task condition was verbalized serial subtractions of 3's. The absolute change was then calculated using post-intervention dual task cost minus baseline dual task cost. Negative numbers demonstrate lower (i.e., better) dual task cost post intervention. The preferred Unit of Measure is unitless.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
unitless | -9.86 (53.03) | -24.96 (27.96) | 4.29 (34.43) | 0.84 (33.18)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task cost to stride time variability from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.04, ANOVA

4. Secondary Outcome: Absolute Change in Single Task Gait Speed From Baseline to Immediately Post Intervention
Description: Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer, on the low back and feet to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed pre and post tDCS. Two at a preferred speed while walking quietly (single task). The absolute change from baseline to immediately post intervention was calculated by averaging the single task gait speeds (m/s) pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m/s | 0.025 (0.01) | 0.031 (0.012) | 0.017 (0.011) | 0.014 (0.012)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized no significant effect of intervention type on absolute change in single task gait speed from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.56, ANOVA

5. Secondary Outcome: Absolute Change in Dual Task Gait Speed From Baseline to Immediately Post Intervention
Description: Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer, on the low back and feet to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed pre and post tDCS. Two at a preferred speed while performing a cognitive task (dual task). The cognitive task during the dual task condition was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change from baseline to immediately post intervention was calculated by averaging the dual task gait speeds (m/s) pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m/s | 0.046 (0.086) | 0.042 (0.048) | -0.002 (0.011) | 0.016 (0.029)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task gait speed from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.07, ANOVA

6. Secondary Outcome: Absolute Change in Single Task Stride Time Variability From Baseline to Immediately Post Intervention
Description: Stride time variability (STV) is a measure of how consistent limb movements are during walking. It's expressed as the coefficient of variation (CoV) and calculated from the mean and standard deviation of stride time. Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer, on the low back and feet to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed. Two at a preferred speed while walking quietly (single task). The absolute change from baseline to immediately post intervention was calculated by averaging the single task stride time variability pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
coefficient of variation | -0.07 (0.09) | -0.04 (0.09) | -0.06 (0.08) | -0.03 (0.09)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized no significant effect of intervention type on absolute change in single task stride time variability from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.74, ANOVA

7. Secondary Outcome: Absolute Change in Dual Task Stride Time Variability From Baseline to Immediately Post Intervention
Description: Stride time variability (STV) is a measure of how consistent limb movements are during walking. It's expressed as the coefficient of variation (CoV) and calculated from the mean and standard deviation of stride time. Prior to testing, participants were outfitted with wireless biosensors, each containing a triaxial accelerometer, goniometer and magnetometer, on the low back and feet to record gait kinematics (Mobility Lab™, APDM Inc). Six 25-meter walking trials were completed. Two at a preferred speed while performing a cognitive task (dual task). The cognitive task during the dual task condition was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change from baseline to immediately post intervention was calculated by averaging the dual task stride time variability pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
coefficient of variation | -0.27 (1.04) | -0.23 (0.37) | -0.16 (0.89) | -0.13 (0.50)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task stride time variability from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.33, ANOVA

8. Secondary Outcome: Absolute Change in Dual Task Cost to Standing Postural Sway Area From Baseline to Immediately Post Intervention
Description: Postural sway area was assessed by measuring postural sway elliptical area during six, 45-second trials of standing with eyes open (single task), eyes closed, or performing a cognitive task (dual task standing) on a stationary force platform (Kistler, Amherst, NY). The cognitive task was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change was then calculated using post-intervention dual task cost minus baseline dual task cost. The outcome was obtained by averaging the dual task costs of the four trials. Negative numbers demonstrate lower (i.e., better) dual task cost post intervention. The preferred Unit of Measure is unitless.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
unitless | -23.17 (82.98) | -3.18 (59.23) | 21.45 (71.17) | -3.23 (58.45)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task cost to standing postural sway area from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.16, ANOVA

9. Secondary Outcome: Absolute Change in Single Task Postural Sway Speed From Baseline to Immediately Post Intervention
Description: Postural sway speed was assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during two, 45-second trials of standing with eyes open (single task) on a stationary force platform (Kistler, Amherst, NY) pre and post intervention. The absolute change from baseline to immediately post intervention was calculated by averaging the single task postural sway speed (m/s) pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m/s | 0.013 (0.023) | -0.018 (0.023) | -0.028 (0.023) | 0.0078 (0.024)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized no significant effect of intervention type on absolute change in single task postural sway speed from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.52, ANOVA

10. Secondary Outcome: Absolute Change in Dual Task Postural Sway Speed From Baseline to Immediately Post Intervention
Description: Postural sway speed was assessed by measuring standing postural sway (ie., center-of pressure fluctuations) during two, 45-second trials of standing with eyes open while performing a cognitive task (dual task) on a stationary force platform (Kistler, Amherst, NY) pre and post intervention. The cognitive task was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change from baseline to immediately post intervention was calculated by averaging the dual task postural sway speed (m/s) pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m/s | -0.0056 (0.016) | -0.0029 (0.018) | 0.063 (0.017) | -0.0001 (0.018)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task postural sway speed from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, ANOVA

11. Secondary Outcome: Absolute Change in Single Task Postural Sway Area From Baseline to Immediately Post Intervention
Description: Postural sway area was assessed by measuring postural sway elliptical area during two, 45-second trials of standing with eyes open (single task) on a stationary force platform (Kistler, Amherst, NY) pre and post intervention. The absolute change from baseline to immediately post intervention was calculated by averaging the single task postural sway area pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m²
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m² | 0.0049 (0.023) | -0.001 (0.021) | 0.0025 (0.012) | 0.01 (0.023)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized no significant effect of intervention type on absolute change in single task postural sway area from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.39, ANOVA

12. Secondary Outcome: Absolute Change in Dual Task Postural Sway Area From Baseline to Immediately Post Intervention
Description: Postural sway area was assessed by measuring postural sway elliptical area during two, 45-second trials of standing with eyes open while performing a cognitive task (dual task) on a stationary force platform (Kistler, Amherst, NY) pre and post intervention. The cognitive task was verbalized serial subtractions of 3's from a random three-digit number between 200 and 999. Participant responses during each trial were recorded. The absolute change from baseline to immediately post intervention was calculated by averaging the dual task postural sway area pre and post.
Time Frame: Change from baseline to immediately post-tDCS, up to 60 minutes
Measure: Mean (Standard Deviation); unit: m²
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
Number analyzed (Participants) | 29 | 29 | 29 | 28
m² | -0.0081 (0.041) | -0.0091 (0.034) | 0.0025 (0.029) | 0.0086 (0.021)
Statistical Analysis 1: Comparison: Conventional tDCS vs Optimized tDCS vs Conventional Sham vs Optimized Sham; We hypothesized a significant effect of intervention type on absolute change in dual task postural sway area from baseline to immediately post intervention; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.18, ANOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Conventional tDCS | Optimized tDCS | Conventional Sham | Optimized Sham
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 1/29 | 1/29 | 3/29 | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional tDCS (N=29) | Optimized tDCS (N=29) | Conventional Sham (N=29) | Optimized Sham (N=28)
Dizziness (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04295798/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04295798/SAP_002.pdf
  • Informed Consent Form (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04295798/ICF_003.pdf